CLINICAL TRIAL: NCT01100073
Title: Kinetic Tremor in Parkinsons Disease: Its Course Under Pramipexole (Mirapexin®) Treatment and Impact on Quality of Life
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 248.657
Record Dates: First submitted 2010-03-18; First posted 2010-04-08 (Estimated); Results first posted 2010-09-20 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with Parkinson's disease: Early and advanced Parkinson's disease patients

SUMMARY:
The study will compare the effect of pramipexole on different types of tremor and particularly kinetic tremor in early and advanced Parkinson's disease patients and will evaluate the course of tremor measured with spiralometry under pramipexole treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic Parkinson's disease with or without fluctuations
2. Indication for treatment with pramipexole (Mirapexin®)
3. Presence of at least mild tremor symptoms (as judged by the treating physician)

Exclusion Criteria:

1. Any contraindications according to the Summary of Product Characteristics (SPC): hypersensitivity to pramipexole or to any of the excipients.
2. Ongoing treatment with pramipexole (Mirapexin®)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Neurologists
Sampling Method: Non-Probability Sample
Enrollment: 1703 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (215):
- Estonia (8):
  - Boehringer Ingelheim Investigational Site 5, Keila
  - Boehringer Ingelheim Investigational Site 4, Kohtla-Järve
  - Boehringer Ingelheim Investigational Site 6, Rakvere
  - Boehringer Ingelheim Investigational Site 1, Tallinn
  - Boehringer Ingelheim Investigational Site 2, Tallinn
  - Boehringer Ingelheim Investigational Site 3, Tallinn
  - Boehringer Ingelheim Investigational Site 7, Tartu
  - Boehringer Ingelheim Investigational Site 8, Valga
- Latvia (23):
  - Boehringer Ingelheim Investigational Site 9, Kuldīga
  - Boehringer Ingelheim Investigational Site 12, Liepāja
  - Boehringer Ingelheim Investigational Site 13, Liepāja
  - Boehringer Ingelheim Investigational Site 14, Liepāja
  - Boehringer Ingelheim Investigational Site 15, Liepāja
  - Boehringer Ingelheim Investigational Site 10, Limbaži
  - Boehringer Ingelheim Investigational Site 11, Limbaži
  - Boehringer Ingelheim Investigational Site 16, Riga
  - Boehringer Ingelheim Investigational Site 17, Riga
  - Boehringer Ingelheim Investigational Site 18, Riga
  - Boehringer Ingelheim Investigational Site 19, Riga
  - Boehringer Ingelheim Investigational Site 20, Riga
  - Boehringer Ingelheim Investigational Site 21, Riga
  - Boehringer Ingelheim Investigational Site 22, Riga
  - Boehringer Ingelheim Investigational Site 23, Riga
  - Boehringer Ingelheim Investigational Site 24, Riga
  - Boehringer Ingelheim Investigational Site 25, Riga
  - Boehringer Ingelheim Investigational Site 26, Riga
  - Boehringer Ingelheim Investigational Site 27, Riga
  - Boehringer Ingelheim Investigational Site 28, Riga
  - Boehringer Ingelheim Investigational Site 29, Riga
  - Boehringer Ingelheim Investigational Site 30, Riga
  - Boehringer Ingelheim Investigational Site 31, Riga
- Romania (93):
  - Boehringer Ingelheim Investigational Site 32, Aiud
  - Boehringer Ingelheim Investigational Site 33, Arges
  - Boehringer Ingelheim Investigational Site 34, Arges
  - Boehringer Ingelheim Investigational Site 35, Arges
  - Boehringer Ingelheim Investigational Site 36, Arges
  - Boehringer Ingelheim Investigational Site 37, Arges
  - Boehringer Ingelheim Investigational Site 38, Arges
  - Boehringer Ingelheim Investigational Site 39, Arges
  - Boehringer Ingelheim Investigational Site 40, Bacau
  - Boehringer Ingelheim Investigational Site 41, Bacau
  - Boehringer Ingelheim Investigational Site 42, Bistriţa
  - Boehringer Ingelheim Investigational Site 43, Botoșani
  - Boehringer Ingelheim Investigational Site 44, Botoșani
  - Boehringer Ingelheim Investigational Site 47, Brasov
  - Boehringer Ingelheim Investigational Site 48, Brasov
  - Boehringer Ingelheim Investigational Site 45, Brăila
  - Boehringer Ingelheim Investigational Site 46, Brăila
  - Boehringer Ingelheim Investigational Site 49, Bucharest
  - Boehringer Ingelheim Investigational Site 50, Bucharest
  - Boehringer Ingelheim Investigational Site 51, Bucharest
  - Boehringer Ingelheim Investigational Site 52, Bucharest
  - Boehringer Ingelheim Investigational Site 53, Bucharest
  - Boehringer Ingelheim Investigational Site 54, Bucharest
  - Boehringer Ingelheim Investigational Site 55, Bucharest
  - Boehringer Ingelheim Investigational Site 56, Bucharest
  - Boehringer Ingelheim Investigational Site 57, Bucharest
  - Boehringer Ingelheim Investigational Site 58, Bucharest
  - Boehringer Ingelheim Investigational Site 59, Bucharest
  - Boehringer Ingelheim Investigational Site 60, Bucharest
  - Boehringer Ingelheim Investigational Site 61, Bucharest
  - Boehringer Ingelheim Investigational Site 62, Bucharest
  - Boehringer Ingelheim Investigational Site 63, Bucharest
  - Boehringer Ingelheim Investigational Site 64, Bucharest
  - Boehringer Ingelheim Investigational Site 65, Bucharest
  - Boehringer Ingelheim Investigational Site 66, Bucharest
  - Boehringer Ingelheim Investigational Site 67, Bucharest
  - Boehringer Ingelheim Investigational Site 68, Bucharest
  - Boehringer Ingelheim Investigational Site 69, Bucharest
  - Boehringer Ingelheim Investigational Site 70, Bucharest
  - Boehringer Ingelheim Investigational Site 71, Bucharest
  - Boehringer Ingelheim Investigational Site 72, Buzău
  - Boehringer Ingelheim Investigational Site 73, Buzău
  - Boehringer Ingelheim Investigational Site 74, Caracal
  - Boehringer Ingelheim Investigational Site 75, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 76, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 77, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 78, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 79, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 80, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 81, Constanța
  - Boehringer Ingelheim Investigational Site 82, Constanța
  - Boehringer Ingelheim Investigational Site 83, Craiova
  - Boehringer Ingelheim Investigational Site 84, Craiova
  - Boehringer Ingelheim Investigational Site 85, Craiova
  - Boehringer Ingelheim Investigational Site 86, Craiova
  - Boehringer Ingelheim Investigational Site 87, Deva
  - Boehringer Ingelheim Investigational Site 88, Deva
  - Boehringer Ingelheim Investigational Site 89, Focşani
  - Boehringer Ingelheim Investigational Site 90, Focşani
  - Boehringer Ingelheim Investigational Site 91, Galati
  - Boehringer Ingelheim Investigational Site 92, Galati
  - Boehringer Ingelheim Investigational Site 93, Hunedoara
  - Boehringer Ingelheim Investigational Site 94, Hunedoara
  - Boehringer Ingelheim Investigational Site 95, Iași
  - Boehringer Ingelheim Investigational Site 96, Iași
  - Boehringer Ingelheim Investigational Site 97, Iași
  - Boehringer Ingelheim Investigational Site 98, Iași
  - Boehringer Ingelheim Investigational Site 99, Lugoj
  - Boehringer Ingelheim Investigational Site 100, Maramures
  - Boehringer Ingelheim Investigational Site 101, Orăştie
  - Boehringer Ingelheim Investigational Site 102, Paşcani
  - Boehringer Ingelheim Investigational Site 103, Paşcani
  - Boehringer Ingelheim Investigational Site 104, Petroşani
  - Boehringer Ingelheim Investigational Site 105, Piatra Neamţ
  - Boehringer Ingelheim Investigational Site 106, Prahova
  - Boehringer Ingelheim Investigational Site 107, Prahova
  - Boehringer Ingelheim Investigational Site 108, Prahova
  - Boehringer Ingelheim Investigational Site 109, Radauti
  - Boehringer Ingelheim Investigational Site 110, Reşiţa
  - Boehringer Ingelheim Investigational Site 111, Satu Mare
  - Boehringer Ingelheim Investigational Site 112, Sibiu
  - Boehringer Ingelheim Investigational Site 113, Sibiu
  - Boehringer Ingelheim Investigational Site 114, Slatina
  - Boehringer Ingelheim Investigational Site 115, Suceava
  - Boehringer Ingelheim Investigational Site 116, Suceava
  - Boehringer Ingelheim Investigational Site 117, Teleorman
  - Boehringer Ingelheim Investigational Site 118, Tg. Mures
  - Boehringer Ingelheim Investigational Site 119, Timișoara
  - Boehringer Ingelheim Investigational Site 120, Timișoara
  - Boehringer Ingelheim Investigational Site 121, Timișoara
  - Boehringer Ingelheim Investigational Site 122, Timișoara
  - Boehringer Ingelheim Investigational Site 123, Tulcea
  - Boehringer Ingelheim Investigational Site 124, Tulcea
- Russia (10):
  - Boehringer Ingelheim Investigational Site 131, Krasnodar
  - Boehringer Ingelheim Investigational Site 130, Krasnoyarsk
  - Boehringer Ingelheim Investigational Site 125, Moscow
  - Boehringer Ingelheim Investigational Site 126, Moscow
  - Boehringer Ingelheim Investigational Site 127, Moscow
  - Boehringer Ingelheim Investigational Site 128, Novosibirsk
  - Boehringer Ingelheim Investigational Site 132, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 133, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 134, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 129, Tomsk
- Serbia (11):
  - Boehringer Ingelheim Investigational Site 135, Belgrade
  - Boehringer Ingelheim Investigational Site 136, Belgrade
  - Boehringer Ingelheim Investigational Site 140, Kragujevac
  - Boehringer Ingelheim Investigational Site 138, Kruševac
  - Boehringer Ingelheim Investigational Site 141, Niš
  - Boehringer Ingelheim Investigational Site 142, Niš
  - Boehringer Ingelheim Investigational Site 137, Novi Sad
  - Boehringer Ingelheim Investigational Site 143, Sombor
  - Boehringer Ingelheim Investigational Site 145, Užice
  - Boehringer Ingelheim Investigational Site 139, Valjevo
  - Boehringer Ingelheim Investigational Site 144, Vranje
- Slovakia (55):
  - Boehringer Ingelheim Investigational Site 155, ?adca
  - Boehringer Ingelheim Investigational Site 146, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 147, Bardejov
  - Boehringer Ingelheim Investigational Site 148, Bratislava
  - Boehringer Ingelheim Investigational Site 149, Bratislava
  - Boehringer Ingelheim Investigational Site 150, Bratislava
  - Boehringer Ingelheim Investigational Site 151, Bratislava
  - Boehringer Ingelheim Investigational Site 152, Bratislava
  - Boehringer Ingelheim Investigational Site 153, Bratislava
  - Boehringer Ingelheim Investigational Site 154, Brezno
  - Boehringer Ingelheim Investigational Site 156, Humenné
  - Boehringer Ingelheim Investigational Site 157, Ilava
  - Boehringer Ingelheim Investigational Site 158, Komárno
  - Boehringer Ingelheim Investigational Site 163, Kosice- Saca
  - Boehringer Ingelheim Investigational Site 159, Košice
  - Boehringer Ingelheim Investigational Site 160, Košice
  - Boehringer Ingelheim Investigational Site 161, Košice
  - Boehringer Ingelheim Investigational Site 162, Košice
  - Boehringer Ingelheim Investigational Site 164, Krompachy
  - Boehringer Ingelheim Investigational Site 165, Levice
  - Boehringer Ingelheim Investigational Site 166, Liptovský Mikulás
  - Boehringer Ingelheim Investigational Site 167, Lučenec
  - Boehringer Ingelheim Investigational Site 168, Martin
  - Boehringer Ingelheim Investigational Site 169, Nitra
  - Boehringer Ingelheim Investigational Site 170, Nitra
  - Boehringer Ingelheim Investigational Site 171, Nitra
  - Boehringer Ingelheim Investigational Site 172, Nováky
  - Boehringer Ingelheim Investigational Site 173, Nové Mesto N/ Váhom
  - Boehringer Ingelheim Investigational Site 174, Pezinok
  - Boehringer Ingelheim Investigational Site 175, Pies?any
  - Boehringer Ingelheim Investigational Site 176, Povazská Bystrica
  - Boehringer Ingelheim Investigational Site 177, Prešov
  - Boehringer Ingelheim Investigational Site 178, Prešov
  - Boehringer Ingelheim Investigational Site 179, Prešov
  - Boehringer Ingelheim Investigational Site 180, Revúca
  - Boehringer Ingelheim Investigational Site 181, Rimavská Sobota
  - Boehringer Ingelheim Investigational Site 182, Rožňava
  - Boehringer Ingelheim Investigational Site 183, Rožňava
  - Boehringer Ingelheim Investigational Site 185, Sereď
  - Boehringer Ingelheim Investigational Site 186, Skalica
  - Boehringer Ingelheim Investigational Site 187, Stropkov
  - Boehringer Ingelheim Investigational Site 184, Šaľa
  - Boehringer Ingelheim Investigational Site 188, Šurany
  - Boehringer Ingelheim Investigational Site 189, Trebišov
  - Boehringer Ingelheim Investigational Site 190, Tren?in
  - Boehringer Ingelheim Investigational Site 191, Trnava
  - Boehringer Ingelheim Investigational Site 192, Trnava
  - Boehringer Ingelheim Investigational Site 193, Trstená
  - Boehringer Ingelheim Investigational Site 194, Veľké Kapušany
  - Boehringer Ingelheim Investigational Site 195, Ziar N/Hronom
  - Boehringer Ingelheim Investigational Site 198, Zlaté Moravce
  - Boehringer Ingelheim Investigational Site 199, Zvolen
  - Boehringer Ingelheim Investigational Site 200, Zvolen
  - Boehringer Ingelheim Investigational Site 196, Žilina
  - Boehringer Ingelheim Investigational Site 197, Žilina
- Slovenia (10):
  - Boehringer Ingelheim Investigational Site 205, Bled
  - Boehringer Ingelheim Investigational Site 206, Celje
  - Boehringer Ingelheim Investigational Site 201, Ljubljana
  - Boehringer Ingelheim Investigational Site 202, Ljubljana
  - Boehringer Ingelheim Investigational Site 207, Maribor
  - Boehringer Ingelheim Investigational Site 208, Maribor
  - Boehringer Ingelheim Investigational Site 209, Maribor
  - Boehringer Ingelheim Investigational Site 210, Maribor
  - Boehringer Ingelheim Investigational Site 203, Šempeter pri Gorici
  - Boehringer Ingelheim Investigational Site 204, Šempeter pri Gorici
- Ukraine (5):
  - Boehringer Ingelheim Investigational Site 212, Kharkiv
  - Boehringer Ingelheim Investigational Site 211, Kyiv
  - Boehringer Ingelheim Investigational Site 215, Lviv
  - Boehringer Ingelheim Investigational Site 214, Ternopil
  - Boehringer Ingelheim Investigational Site 213, Vinnitsa

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: * enrolled in study: 1703
  * treated (received Mirapexin): 1699 (i.e. 4 patients no record of receiving treatment)
  * completed study: 1599 (i.e. 100 discontinued prematurely)
Groups:
- Mirapexin® (Pramipexole): Mirapexin® (Pramipexole) - tablets for oral use. The dose of Mirapexin® was selected by the treating physician upon his/her clinical judgement and on individual patient need, according to recommendations given in the Mirapexin® Summary of Product Characteristics.
Period: Overall Study
Arm/Group | Mirapexin® (Pramipexole)
Started | 1699 (Baseline (Visit 1))
Completed | 1599 (End of study (Visit 3))
Not Completed | 100
Not completed — Lack of Efficacy | 4
Not completed — Insufficient Tolerability | 21
Not completed — Withdrawal by Subject | 13
Not completed — Lost to Follow-up | 39
Not completed — Lack of effect + patient's wish | 2
Not completed — Insufficient tolerability +patients wish | 8
Not completed — Other | 8
Not completed — Missing | 5

BASELINE CHARACTERISTICS:
Population: Treated set (TS) (31 patients were missing age and 17 patients were missing gender)
Groups:
- Mirapexin® (Pramipexole): Mirapexin® (Pramipexole) - tablets for oral use The dose of Mirapexin® was selected by the treating physician upon his/her clinical judgement and on individual patient need, according to recommendations given in the Mirapexin® Summary of Product Characteristics.
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 1699
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (9.70)
Sex/Gender, Customized [Number; unit: participants]
  Female | 844
  Male | 838
  Category title missing | 17

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part II Score at the End of Maintenance
Description: Change (reduction) in UPDRS Part II score (activities of daily living) from baseline to end of study. Score ranging from 0 - 52 (0=no disability, 52=maximum disability)
Time Frame: Week 0 to weeks 9-16 (Visit 3)
Population: Full analysis set (FAS) - Patients for whom baseline and end of study UPDRS Part II scores available
Measure: Mean (Standard Deviation); unit: Points on UPDRS scale
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 1424
Points on UPDRS scale | 5.20 (4.5)

2. Primary Outcome: Change From Baseline in UPDRS Part III Score at the End of Maintenance
Description: Change (reduction) in UPDRS Part III score (motor function) from baseline to end of study. Score ranging from 0 - 108 (0=no disability, 108=maximum disability)
Time Frame: Week 0 to weeks 9-16
Population: Full analysis set (FAS) - Patients for whom baseline and end of study UPDRS Part III scores available
Measure: Mean (Standard Deviation); unit: Points on UPDRS scale
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 1094
Points on UPDRS scale | 12 (9.9)

3. Primary Outcome: Change From Baseline in Spiralometry Measurement at the End of Maintenance (Right Hand)
Description: Change (reduction) in tremor amplitude from baseline to end of study for the right hand
Time Frame: Week 0 to weeks 9-16 (Visit 3)
Population: Full analysis set (FAS) - Patients for whom baseline and end of study spiralometry measurement (right hand) available
Measure: Mean (Standard Deviation); unit: millimeters of tremor amplitude
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 949
millimeters of tremor amplitude | 0.3 (1.6)

4. Primary Outcome: Change From Baseline in Spiralometry Measurement at the End of Maintenance (Left Hand)
Description: Change (reduction) in tremor amplitude from baseline to end of study for the left hand
Time Frame: Week 0 to weeks 9-16 (Visit 3)
Population: Full analysis set (FAS) - Patients for whom baseline and end of study spiralometry measurement (left hand) available
Measure: Mean (Standard Deviation); unit: millimeters of tremor amplitude
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 962
millimeters of tremor amplitude | 0.2 (1.7)

5. Primary Outcome: Change From Baseline in Tremor Score From UPDRS (Items 16, 20, 21) at the End of Maintenance (Visit 3)
Description: Change (reduction)in tremor score from baseline to end of study. Score ranging from 0 - 32 (0=no tremor, 32=high tremor)
Time Frame: Week 0 to weeks 9-16 (Visit 3)
Population: Full analysis set (FAS) - Patients for whom baseline and end of study UPDRS tremor score (UPDRS items 16, 20, 21) available
Measure: Mean (Standard Deviation); unit: Points on UPDRS scale
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 1169
Points on UPDRS scale | 4.1 (3.4)

6. Primary Outcome: Change From Baseline in 39 Item Parkinson's Disease Questionnaire (PDQ-39) Score at the End of Maintenance
Description: Change (reduction) in PDQ-39 score (quality of life) from baseline to end of study. Score ranging from 0-100 (0=perfect health, 100=worst health as assessed by the measure)
Time Frame: Week 0 to weeks 9-16 (Visit 3)
Population: Full analysis set (FAS) - Patients for whom baseline and end of study PDQ-39 score available
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 1239
unit on a scale | 15 (18.4)

7. Secondary Outcome: Final Dose Distribution
Description: Final Mirapexin® dose distribution at the end of study
Time Frame: Enter Week 0 to weeks 9-16 (Visit 3)
Population: Total patients. Number of participants analysed differs for each outcome measure because not all evaluations were performed / documented on every patient.
Measure: Median (Full Range); unit: milligrams of Mirapexin® (salt)
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 1623
milligrams of Mirapexin® (salt) | 3.0 [0.25 to 7.5]

8. Secondary Outcome: Change From Baseline in UPDRS Part II Score at the End of Up-titration
Description: Change (reduction) in UPDRS Part II score (activities of daily living) from baseline to Visit 2. Score ranging from 0 - 52 (0=no disability, 52=maximum disability)
Time Frame: Enter Week 0 to weeks 1-8 (Visit 2)
Population: Patients for whom baseline and Visit 2 UPDRS Part II scores available
Measure: Mean (Standard Deviation); unit: Points on a UPDRS scale
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 1490
Points on a UPDRS scale | 3.1 (3.5)

9. Secondary Outcome: Change From Baseline in UPDRS Part III Score at the End of Up-titration
Description: Change (reduction) in UPDRS Part III score (motor function) from baseline to Visit 2. Score ranging from 0 - 108 (0=no disability, 108=maximum disability)
Time Frame: Enter Week 0 to weeks 1-8 (Visit 2)
Population: Patients for whom baseline and Visit 2 UPDRS Part III scores available
Measure: Mean (Standard Deviation); unit: Points on a UPDRS scale
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 1131
Points on a UPDRS scale | 7.6 (8.1)

10. Secondary Outcome: Change in Tremor Score (UPDRS Items 16, 20, 21) at the End of Up-titration
Description: Change (reduction) from baseline in tremor score, derived from UPDRS from baseline to Visit 2. Score ranging from 0 - 32 (0=no tremor, 32=high tremor)
Time Frame: Enter Week 0 to weeks 1-8 (Visit 2)
Population: Patients for whom baseline and Visit 2 UPDRS Part II and III scores available
Measure: Mean (Standard Deviation); unit: Points on a UPDRS scale
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 1207
Points on a UPDRS scale | 2.5 (2.9)

11. Secondary Outcome: Incidence, Relationship and Seriousness of Adverse Events
Description: Total number of adverse events (AEs), causality and level of seriousness
Time Frame: Week 0 to weeks 9-16 (end of study)
Population: Total patients
Measure: Number; unit: Number of events
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 1699
Number of events
  Incidence (Total number of AEs) | 266
  Related (Number of treatment related AEs) | 230
  SAE (Number of serious adverse events) | 3

12. Secondary Outcome: Number of Premature Discontinuations
Description: Number of patients discontinuing the study prematurely
Time Frame: Week 0 to weeks 9-16 (end of study)
Population: Total patients
Measure: Number; unit: Participants
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 1699
Participants | 100

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Arm/Group | Mirapexin® (Pramipexole)
Serious Adverse Events (participants affected / at risk) | 3/1699
Other Adverse Events (participants affected / at risk) | 0/1699
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirapexin® (Pramipexole) (N=1699)
Vertebral Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute Stroke (Nervous system disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract